CLINICAL TRIAL: NCT04818229
Title: A Phase I, Multicenter, Randomized, Double-blind, Double-dummy, Placebo- and Positive-Controlled Study to Investigate the Effects of CBP-307 on the QTc Interval in Healthy Subjects
Brief Title: A Study to Investigate the Effects of CBP-307 on the Heart Rate-corrected QT Interval (QTc) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connect Biopharma Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Connect Biopharm LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CBP-307AU002
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Group 1 (Experimental): Therapeutic and supratherapeutic multiple oral doses of CBP-307.
  Interventions: Drug: CBP-307; Drug: Placebo-matched CBP-307
- Investigational Group 2A (Placebo Comparator): Moxifloxacin (positive control for method validation) and Placebo oral administration.
  Interventions: Drug: Moxifloxacin (Avelox); Drug: Placebo-matched Moxifloxacin
- Investigational Group 2B (Placebo Comparator): Moxifloxacin (positive control for method validation) and Placebo oral administration.
  Interventions: Drug: Moxifloxacin (Avelox); Drug: Placebo-matched Moxifloxacin

INTERVENTIONS:
Drug: CBP-307 — CBP-307 capsules oral administration.
  Arms: Investigational Group 1
Drug: Placebo-matched CBP-307 — Placebo-matched CBP-307 capsules oral administration.
  Arms: Investigational Group 1
Drug: Moxifloxacin (Avelox) — Moxifloxacin tablets oral administration。
  Arms: Investigational Group 2A; Investigational Group 2B
Drug: Placebo-matched Moxifloxacin — Placebo-matched Moxifloxacin tablets oral administration.
  Arms: Investigational Group 2A; Investigational Group 2B

SUMMARY:
This study will investigate the effects of therapeutic and supratherapeutic oral doses of CBP-307 on the QTc interval in healthy subjects.

DETAILED DESCRIPTION:
This will be a Phase I, randomized, double-blind, double-dummy, placebo-controlled, positive-controlled, multi-site, 3-arm study to investigate the effects of therapeutic and supratherapeutic oral doses of CBP-307 on the QTc interval in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 60 years of age, inclusive.
2. Body mass index between 18.0 and 30.0 kg/mE2, inclusive.
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and confirmed at check-in as assessed by the investigator (or designee).
4. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception. Negative pregnancy test for females of childbearing potential at screening (blood test) and check-in (urine test).
5. Supine diastolic blood pressure between 60 and 90 mmHg and systolic blood pressure between 90 and 140 mmHg (inclusive) at screening on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
6. No clinically significant history or presence of ECG findings as judged by the investigator at screening and check-in, including each criterion as listed below:

   1. Normal sinus rhythm (HR between 55 bpm and 100 bpm inclusive);
   2. QTcF interval ≤450 msec for males and females;
   3. QRS interval ≤110 msec; and confirmed by manual over-read if >110 msec;
   4. PR interval ≤200 msec.
7. Has serum potassium, calcium, and magnesium levels within the normal reference range at screening, as judged by the investigator.
8. Able to swallow multiple tablets (based on subject's verbal confirmation).
9. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.

Exclusion Criteria:

-

Subjects will be excluded from the study if they satisfy any of the following criteria at the screening visit unless otherwise stated:

1. Subject is mentally or legally incapacitated or has had significant history of recent mental health issues requiring medication and/or hospitalization at the time of the screening visit or expected during the conduct of the study.
2. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee). Note: Childhood asthma that is considered recovered or seasonal allergies that are not currently active or requiring treatment are allowed.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
4. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs, related compounds, or inactive ingredients.
5. History of significant multiple and/or severe allergies (eg, latex allergy, band-aids, adhesive dressing, or medical tape), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs.
6. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs within 6 months prior to the first dose of study drug (uncomplicated appendectomy and hernia repair will be allowed).
7. History or presence of:

   1. Hypokalemia, in the opinion of the investigator (or designee);
   2. Risk factors for Torsades de Pointes (eg, heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   3. Sick sinus syndrome, second, or third degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities;
   4. Repeated or frequent syncope or vasovagal episodes;
   5. Hypertension, angina, bradycardia, or severe peripheral arterial circulatory disorders.
8. Clinically significant abnormalities (as judged by the investigator in laboratory tests results [out-of-range results confirmed on repeat]), including but not limited to the following parameters:

   1. alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or total bilirubin greater than 1.5 × upper limit of normal;
   2. hemoglobin <10 g/dL, WBC <3.0 ×10E9/L, neutrophils <1.5 ×10E9/L, lymphocytes <0.8 ×10E9/L and platelets <100 ×10E9/L or >1200 × 10E9/L;
9. History or evidence of alcoholism or drug/chemical abuse within 2 years prior to check-in.
10. Alcohol consumption of >10 units per week for males and females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
11. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at screening or check-in.
12. Positive hepatitis panel, positive syphilis test, and/or positive human immunodeficiency virus test.
13. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 28 days prior to the first dose of study treatment on Day 1. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
14. Participation in a previous clinical study where subjects received CBP-307.
15. Administration of a Coronavirus Disease 2019 (COVID-19) vaccine in the past 28 days prior to first dose of study treatment on Day 1.
16. Use or intend to use any prescription medications/products within 14 days prior to first dose of study drug (Day 1) and throughout the study, unless deemed acceptable by the investigator (or designee). Note: For females only, the use hormonal contraception, hormone replacement therapy or oral, implantable, transdermal, injectable, or intrauterine hormonal contraceptives within 14 days prior to Day 1 is not acceptable, except for Mirena®.
17. Use or intend to use any drugs known to be significant inhibitors or inducers of CYP enzymes and/or P-gp, including St. John's Wort, for days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the investigator or designee to confirm the lack of PK/PD interaction with the study drug.
18. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
19. Use or intend to use any nonprescription medications/products including antacids, vitamins (especially those containing magnesium, aluminum, iron, or zinc), minerals, and phytotherapeutic/herbal/plant-derived preparations within 14 days prior to check-in, unless deemed acceptable by the investigator (or designee).
20. Use of tobacco- or nicotine-containing products within 3 months prior to check-in, or positive cotinine at screening or check-in.
21. Has been on a diet incompatible with the on-study diet (including an extreme diet which resulted in a significant weight change for whatever reason), in the opinion of the investigator, within the 28 days prior to the first dose of study treatment, and throughout the study.
22. Consumption of caffeine/xanthine-containing foods or beverages within 48 hours prior to check-in until discharge.
23. Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to check-in.
24. Receipt of blood products within 2 months prior to check-in.
25. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
26. Poor peripheral venous access.
27. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Australia Connect, Study Director — Connect Biopharma Australia Pty Ltd; Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (2):
- Clinical Pharmacology of Miami (CPMI), LLC, Hialeah, Florida, United States
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Placebo was administered to all subjects on Day -1, and assigned study treatments were administered on Days 1 through 16.
Groups:
- Investigational Group 1: In Group 1, subjects received a starting dose of 0.05 mg CBP-307 on Day 1 followed by an up-titrated dose of 0.1 mg on Day 2 and a dose of 0.2 mg on Days 3 to 6 in order to achieve a therapeutic dose on Day 6. Dose administration continued with a dose of 0.5 mg CBP-307 on Days 7 to 15 in order to achieve a supratherapeutic dose on Day 15. CBP-307 and moxifloxacin placebo were administered on Day 16.
- Investigational Group 2A: In Group 2A, 400 mg moxifloxacin was administered on Day 1, with CBP-307 or moxifloxacin placebo administered on all other days.
- Investigational Group 2B: In Group 2B, 400 mg moxifloxacin was administered on Day 16, with CBP-307 or moxifloxacin placebo administered on all other days.
Period: Overall Study
Arm/Group | Investigational Group 1 | Investigational Group 2A | Investigational Group 2B
Started | 55 | 28 | 29
Completed | 32 | 17 | 15
Not Completed | 23 | 11 | 14
Not completed — The cohort was canceled due to COVID-19 | 20 | 10 | 10
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Group 1 | Investigational Group 2A | Investigational Group 2B | Total
Number analyzed (Participants) | 55 | 28 | 29 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (11.17) | 41.6 (11.25) | 41.1 (11.10) | 41.6 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 13 | 11 | 47
  Male | 32 | 15 | 18 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 22 | 23 | 90
  Not Hispanic or Latino | 10 | 6 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 4 | 2 | 15
  White | 45 | 23 | 25 | 93
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 169.13 (10.712) | 168.45 (8.960) | 168.14 (9.821) | 168.71 (9.994)
Body Weight [Mean (Standard Deviation); unit: Kg] | 76.80 (12.481) | 76.70 (10.636) | 76.39 (10.890) | 76.67 (11.543)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.74 (2.656) | 26.95 (2.423) | 27.01 (2.866) | 26.87 (2.636)

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline QT Interval Corrected for Heart Rate Using Fridericia's Method (QTcF)
Description: Change from Baseline in QT interval corrected for heart rate using Fridericia's method (QTcF) to evaluate the effects of therapeutic and supratherapeutic CBP-307 plasma concentrations.
Time Frame: From Baseline to Day 16
Population: Per protocol, approximately 68 healthy subjects (at least 30% for each sex) will be randomized into 2 groups (Group 1 and 2) with 34 subjects in each. Group 2 consists of 2 sub-groups (Group 2A and 2B) and each sub-group will be randomized with 17 subjects. That is to say, the placebo group is consist of Group 2A+Group 2B. The aim is to assess the ECG effect of CBP-307 versus placebo (CBP-307 in Group 1 versus placebo in Groups 2A and 2B).
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Investigational Group 1: 0.5 mg CBP-307 on Day 15 at 24 hours Post-dose.
- Investigational Group 2A+2B: Placebo on Day 15 at 24 hours Post-dose.
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 33
msec | 1.5 (2.46) | 0.9 (2.40)

2. Secondary Outcome: Change-from-baseline Heart Rate (HR)
Description: Change from Baseline in heart rate (HR).
Time Frame: From Baseline at Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats/min
Groups:
- Investigational Group 1: 0.5mg CBP-307 on Day 15 at 24 hours post-dose.
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 33
beats/min | -3.2 (0.98) | -1.3 (0.96)

3. Secondary Outcome: Change-from-baseline PR
Description: Change from Baseline in PR.
Time Frame: From Baseline at Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Groups:
- Investigational Group 2A+2B: Placebo on Day15 at 24 hours Post-dose.
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 33
msec | 4.5 (2.58) | -0.3 (2.51)

4. Secondary Outcome: Change-from-baseline QRS
Description: Change from Baseline in QRS.
Time Frame: From Baseline at Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 33
msec | 0.1 (0.84) | -0.5 (0.81)

5. Secondary Outcome: Placebo-corrected Change-from-baseline HR
Description: Placebo-corrected Change-from-baseline HR based on Change-from-baseline Heart Rate (HR) reported in Outcome Measure 2
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 32
beats/min | -1.9 (1.37)

6. Secondary Outcome: Placebo-corrected Change-from-baseline QTcF
Description: Placebo-corrected change-from-baseline QT Interval Corrected for Heart Rate Using Fridericia's Method (QTcF) based on Change-from-baseline QTcF reported in Outcome Measure 1
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 32
msec | 0.6 (3.44)

7. Secondary Outcome: Placebo-corrected Change-from-baseline PR
Description: Placebo-corrected change-from-baseline PR based on Change-from-baseline PR reported in Outcome Measure 3
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 32
msec | 4.8 (3.60)

8. Secondary Outcome: Placebo-corrected Change-from-baseline QRS
Description: Placebo-corrected change-from-baseline QRS based on Change-from-baseline QRS reported in Outcome Measure 4
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 32
msec | 0.6 (1.17)

9. Secondary Outcome: Categorical Outliers for QTcF
Description: For categorical outliers, the number (percentage) of subjects as well as timepoints who had increases in absolute QTcF values >450 and ≤480 msec, >480 and ≤500 msec, or >500 msec, and changes from predose baseline of >30 and ≤60 msec, or >60 msec.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Investigational Group 1: 0.5mg CBP-307 from Baseline to Day 16
- Investigational Group 2A+2B: Placebo from Baseline to Day 16
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants
  QTcF >450 and ≤480 msec | 1 | 3
  QTcF > 480 and ≤500 ms | 0 | 0
  QTcF > 500 ms | 0 | 0
  Change-from-baseline QTcF >30 and ≤60 ms | 1 | 2
  Change-from-baseline QTcF >60 ms | 0 | 1

10. Secondary Outcome: Categorical Outliers for HR
Description: For categorical outliers, decrease in HR from predose baseline >25% to an HR <50 bpm will be determined.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants | 0 | 1

11. Secondary Outcome: Categorical Outliers for PR
Description: For categorical outliers, increase in PR from predose baseline >25% to a PR > 200 msec will be determined.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants | 0 | 0

12. Secondary Outcome: Categorical Outliers for QRS
Description: For categorical outliers, increase in QRS from predose baseline >25% to a QRS >120 msec will be determined.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants | 0 | 0

13. Secondary Outcome: Frequency of Treatment-emergent Changes of T-wave Morphology
Description: For T-wave morphology, the analyses will be focused on change from baseline with counts (percentages) for both the number of subjects and the number of timepoints.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants
  Flat | 0 | 2
  Notched (+) | 0 | 0
  Biphasic | 0 | 2
  Normal (-) | 0 | 0
  Notched (-) | 0 | 0
  Inverted | 1 | 9

14. Secondary Outcome: Frequency of Treatment-emergent Changes of U-wave Presence
Description: For U-wave presence, the analyses will be focused on change from baseline with counts (percentages) for both the number of subjects and the number of timepoints.
Time Frame: From Baseline to Day 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Group 1 | Investigational Group 2A+2B
Number analyzed (Participants) | 32 | 56
Participants | 0 | 0

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf)
Description: Area under the concentration-time curve from time zero extrapolated to infinity (AUCinf) will be analyzed as a pharmacokinetic (PK) parameter.
Time Frame: From Baseline to Day 29 ± 2
Population: Only subjects in Group 1 received CBP-307.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Investigational Group 1: 0.5mg CBP-307 on Day 15
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 44
h*ng/mL | 543 (24.4)

16. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC0-24)
Description: Area under the concentration-time curve from time zero to 24 hours postdose (AUC0-24) will be analyzed as a pharmacokinetic (PK) parameter.
Time Frame: From Baseline to Day 29 ± 2
Population: Only subjects in Group 1 received CBP-307.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 44
h*ng/mL | 237 (21.8)

17. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration (Cmax) will be analyzed as a pharmacokinetic (PK) parameter.
Time Frame: From Baseline to Day 29 ± 2
Population: Only subjects in Group 1 received CBP-307.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 44
ng/mL | 13.5 (22.0)

18. Secondary Outcome: Time of the Maximum Observed Concentration (Tmax)
Description: Time of the maximum observed concentration (tmax) will be analyzed as a pharmacokinetic (PK) parameter.
Time Frame: From Baseline to Day 29 ± 2
Population: Only subjects in Group 1 received CBP-307.
Measure: Median (Full Range); unit: h
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 44
h | 3.02 [1.02 to 8.00]

19. Secondary Outcome: Incidence and Severity of Adverse Event (AE)
Description: All AEs will be listed and treatment-emergent AEs will be summarized using the descriptive methodology.
  14.3.1.1 TEAE
Time Frame: From Baseline to Day 29 ± 2
Population: Only subjects in Group 1 received CBP-307.
Measure: Number; unit: participants
Arm/Group | Investigational Group 1
Number analyzed (Participants) | 50
participants
  Overall | 12
  Serious | 0
  Leading to Discontinuation | 1
  Leading to Death | 0

ADVERSE EVENTS:
Time Frame: Both AEs and SAEs were recorded from the time the patient signs the ICF (28 days before Day 1) until the follow-up visit (Day 29±2 days) or at early termination. The longest period of time over which adverse event data were collected is 59 days.
Description: Safety outcome measures included incidence and severity of adverse events, incidence of laboratory abnormalities, 12-lead ECG parameters, and vital sign measurements. Per protocol, approximately 68 healthy subjects will be randomized into 2 groups (Group 1 and 2). Only subjects in Group 1 received CBP-307, while all subjects in Group2 received CBP-307 matched placebo. When evaluating the safety of CBP-307 in this study, using combined Group 2 (Group 2A and 2B) as control group is reasonable.
Groups:
- 0.05 mg CBP-307: 0.05 mg CBP-307 on Day 1
- 0.1 mg CBP-307: 0.1 mg on Day 2
- 0.2 mg CBP-307: 0.2 mg on Days 3 to 6
- 0.5 mg CBP-307: 0.5 mg CBP-307 on Days 7 to 15
- Investigational Group 2A+2B: Moxifloxacin (positive control for method validation) and Placebo oral administration.
  Moxifloxacin (Avelox): Moxifloxacin tablets oral administration。
  Placebo-matched Moxifloxacin: Placebo-matched Moxifloxacin tablets oral administration.
Arm/Group | 0.05 mg CBP-307 | 0.1 mg CBP-307 | 0.2 mg CBP-307 | 0.5 mg CBP-307 | Investigational Group 1 | Investigational Group 2A+2B
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/50 | 0/55 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/55 | 0/50 | 0/55 | 0/57
Other Adverse Events (participants affected / at risk) | 4/55 | 7/55 | 14/55 | 12/50 | 22/55 | 22/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.05 mg CBP-307 (N=55) | 0.1 mg CBP-307 (N=55) | 0.2 mg CBP-307 (N=55) | 0.5 mg CBP-307 (N=50) | Investigational Group 1 (N=55) | Investigational Group 2A+2B (N=57)
COVID-19 (Infections and infestations) | 0 | 0 | 4 | 5 | 9 | 11
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 4
Catheter site bruise (General disorders) | 1 | 0 | 0 | 1 | 2 | 1
Medical device site dermatitis (General disorders) | 0 | 1 | 0 | 0 | 1 | 2
Catheter site irritation (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Medical device site irritation (General disorders) | 0 | 1 | 0 | 0 | 1 | 1
Medical device site pruritus (General disorders) | 2 | 0 | 0 | 0 | 2 | 0
Medical device site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 2 | 0
Application site vesicles (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Medical device site erythema (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 4
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 4 | 0 | 4 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ear discomfort (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04818229/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04818229/SAP_001.pdf